CLINICAL TRIAL: NCT05620212
Title: Investigating the Meaning and (Cost-)Effectiveness of Dutch Recovery Colleges
Status: Completed | Type: Observational
Sponsor: Tilburg University (Other)
Collaborators: Trimbos-institute (also primary organization conducting the study) (Unknown); Lister (Unknown); Gemeente Utrecht (Unknown); Stichting tot steun VCVGZ (Other)
Responsible Party: Principal Investigator, Hans Kroon, PhD, Tilburg University
Other Study IDs: TSB_RP390
Record Dates: First submitted 2022-10-27; First posted 2022-11-17 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Severe Mental Illness; Mental Vulnerabilities
Keywords: Recovery Colleges; Empowerment; Severe Mental Illness; Recovery; Effectiveness; Cost-effectiveness
MeSH Terms: conditions — Mental Disorders; Empowerment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RC Group: Recovery College partakers in any way (see description of intervention).
  Interventions: Behavioral: Recovery College participation
- Control Group: Participants with similar mental health profile as RC group, but do not participate in an RC. These participants are sampled from the Panel Psychisch Gezien (PPG), monitored by the Trimbos-institute.

INTERVENTIONS:
Behavioral: Recovery College participation — Recovery College participation in any way (visitors, course/retreat participants, volunteers, employees).
  Groups: RC Group

SUMMARY:
Recovery colleges (RC) aim to promote the recovery of people who experience mental vulnerabilities. Rather than facilitating treatment of illness (as regular mental health care services [MHCS] do), RCs are learning environments, with a special focus on peer support and co-creation. While MHCS are founded on scientific and professional knowledge, RCs value the knowledge and abilities of those with lived experiences as such. By sharing experiences, RC attendees can inspire and support each other (hence 'peer support') and they can use their experiences to contribute to the educational program (hence 'co-creation'). In the Netherlands RCs are 100% peer run, meaning that no mental health care workers are involved.

Despite promising premature findings on the effectiveness of RC attendance (e.g., positive impacts on MHCS use, mental wellbeing and functioning, quality of life, empowerment and more), large, controlled studies are extremely scarce. Furthermore, the way RCs are managed in the Netherlands seems to differ from the RCs that have been studied before. While RCs in some countries are a coproduction of peers and mental health practitioners, RCs in the Netherlands are 100% peer run, although they are usually hosted by MHCS. In turn, this research project aims to investigate the (cost-)effectiveness of RCs in the Netherlands. In terms of effectiveness, we expect that RC attendance improves feelings of empowerment. Besides, we investigate impacts on quality of life, mental health, loneliness, satisfaction with treatment and support and self-stigma. We also determine the cost-effectiveness of Dutch RCs.

DETAILED DESCRIPTION:
This quantitative study is part of a larger research project that entails qualitative analysis of:

* the meaning of Enik RC for its partakers (the first RC established in the Netherlands in 2015);
* the position that RCs can and should have in the Dutch MHCS landscape;
* a fidelity measure to define the core elements of Dutch RCs and to obtain an overview of the available initiatives in the Netherlands

The research project is executed in close collaboration with co-researchers who are partakers of Enik RC. The findings of the pre-registered quantitative study will be evaluated and contextualized in co-creation as such.

NOTE: The Observational Study Model is both Cohort (monitoring for a period of 2 years) and Case-Control (comparing RC partakers with non-partakers).

NOTE: Enik Recovery College has 7 established locations in the region of Utrecht at the time of our recruitment. All are included.

NOTE: Fameus has 4 established locations (Breda 2x, Tilburg, Roosendaal). All are included.

NOTE: This study is conducted both by Tilburg University (Department Tranzo) and Trimbos-institute (Department of Reintegration and Community Care) as primary organizations. The PI is also affiliated with both.

NOTE. The aimed sample size at t0 is N=120 in the RC condition. So 120 partakers of RCs will be matched with members from the PPG.

ELIGIBILITY:
Inclusion Criteria:

* For RC group: needs to attend one of the four participating RCs regularly, at least more than once.
* Needs to experience severe mental illness/psychological vulnerabilities (both self-reported or officially diagnosed).
* Needs to master the Dutch language to sufficient extent to understand the surveys.
* Is 18 years or older.

Exclusion Criteria:

* For the RC group: does not attend one of the four participating RCs regularly.
* Does not experience severe mental illness/psychological vulnerabilities.
* Does not master the Dutch language to a sufficient extent.
* Is younger than 18 years old.
* For the control group (PPG): attends an RC regularly, but not one of the four participating RCs. If an existing PPG member attends one of the four participating RCs regularly, they are allocated to the RC group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RC population (RC Group): Partakers in any way from these four Recovery Colleges: Enik Recovery College, Fameus, Korak, Herstelacademie Haarlem en Meer.
  PPG population (Control Group): National panel for which participants are recruited via mental health care facilities and Regional Institutes for Protected Living (RIPLs).
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Empowerment | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of four subscales (Confidence and Purpose, Connectedness, Self-management and Professional help) of the Netherlands Empowerment List.
  Source: Boevink, W., Kroon, H., Delespaul, P., & Van Os, J. (2016). Empowerment according to persons with severe mental illness: development of the Netherlands empowerment list and its psychometric properties. Open Journal of Psychiatry, 7(1), 18-30. http://dx.doi.org/10.4236/ojpsych.2017.71002

SECONDARY OUTCOMES:
Change in Quality of Life (effectiveness) | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of the Maastricht QoL Scale. Source: Drukker, M., Bak, M., à Campo, J., Driessen, G., Van Os, J., & Delespaul, P. (2010). The cumulative needs for care monitor: a unique monitoring system in the south of the Netherlands. Social psychiatry and psychiatric epidemiology, 45(4), 475-485. https://link.springer.com/content/pdf/10.1007/s00127-009-0088-3.pdf
Change in Mental Health (effectiveness) | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of the MHI-5 scale. Source: Rumpf, H. J., Meyer, C., Hapke, U., & John, U. (2001). Screening for mental health: validity of the MHI-5 using DSM-IV Axis I psychiatric disorders as gold standard. Psychiatry research, 105(3), 243-253. https://doi.org/10.1016/S0165-1781(01)00329-8
Change in Loneliness (effectiveness) | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of the DeJong Gierveld Loneliness Scale. Source: De Jong-Gierveld, J., & Van Tilburg, T. (1990). Manual of the loneliness scale. Amsterdam, Netherlands: Vrije Universiteit.
Change in Satisfaction with Treatment and Support (effectiveness) | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of an inventory adapted from Nivel. Source: Menting, J. De Zorgmonitor - Nationaal Panel Chronisch zieken en Gehandicapten. Uit: www.nivel.nl [Laatst gewijzigd op 18-03-2021; geraadpleegd op 30-08-2022]. URL: https://www.nivel.nl/nl/nationaal-panel-chronisch-zieken-en-gehandicapten/de-zorgmonitor
Change in Self-stigma (effectiveness) | t0 = baseline, t1= 1 year later, t2 = 2 years later.
  Operationalized by means of the ISMI-10 scale. Source: Boyd, J. E., Otilingam, P. G., & DeForge, B. R. (2014). Brief version of the Internalized Stigma of Mental Illness (ISMI) scale: Psychometric properties and relationship to depression, self esteem, recovery orientation, empowerment, and perceived devaluation and discrimination. Psychiatric Rehabilitation Journal, 37(1), 17-23. https://doi.org/10.1037/prj0000035

OTHER OUTCOMES:
Change Health Care and Services Use (cost-effectiveness) | t0 = baseline, t1= 0.5 year later, t2 = 1 year later, t3 = 1.5 years later, t4 = 2 years later.
  Use of health care facilities (e.g., GP, mental health care facilities, psychiatric hospital), services use (e.g., municipality services) and medication, to be transformed into economic costs by the use of the iMTA costing tool.
  Source: Kanters TA, Bouwmans CAM, Van der Linden N, Tan SS, Hakkaart-van Roijen L. Update of the Dutch manual for costing studies in health care. Plos One.
Change in Health Status (cost-effectiveness) | t0 = baseline, t1= 0.5 year later, t2 = 1 year later, t3 = 1.5 years later, t4 = 2 years later.
  Operationalized by means of the EQ-5D. Source: Rabin, R., & Charro, F. D. (2001). EQ-SD: a measure of health status from the EuroQol Group. Annals of medicine, 33(5), 337-343. https://doi.org/10.3109/07853890109002087
Change in Employment Status (cost-effectiveness) | t0 = baseline, t1= 0.5 year later, t2 = 1 year later, t3 = 1.5 years later, t4 = 2 years later.
  Whether or not the participant has paid employment or a volunteering job.
Change in Absenteeism and Presenteeism (cost-effectiveness) | t0 = baseline, t1= 0.5 year later, t2 = 1 year later, t3 = 1.5 years later, t4 = 2 years later.
  The amount of working days participants were ill and could not work (absenteeism), and the amount of working days participants were ill but still went to work (presenteeism). Regarding presenteeism we inquire about the % of work done as compared to an average working day. This will be transformed into costs.
Change in Providing and Receiving Informal Care (cost-effectiveness) | t0 = baseline, t1= 0.5 year later, t2 = 1 year later, t3 = 1.5 years later, t4 = 2 years later.
  Questions whether participant provides informal care (and if so, how many hours per week) and whether participant receives informal care from e.g., family or friends (and if so, how many hours per week). This will be transformed into costs.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Korak, Apeldoorn
  - Herstelacademie Haarlem en Meer, Haarlem
  - Fameus, Tilburg
  - Enik Recovery College, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Upon request.
Access Criteria: PI reviews requests.

REFERENCES:
- [Derived] van Wezel MMC, Muusse C, van de Mheen D, Wijnen B, den Hollander W, Kroon H. What do we not know (yet) about recovery colleges? A study protocol on their (cost-)effectiveness, mechanisms of action, fidelity and positioning. BMC Psychiatry. 2023 Nov 8;23(1):816. doi: 10.1186/s12888-023-05293-8. PMID 37940915